CLINICAL TRIAL: NCT03254121
Title: Genome Studies of Hepatocellular Carcinoma Developed in Hepatitis C Patients With Sustained Virological Response
Acronym: HEPCASUS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Soo Aleman, MD, PhD, Assoc prof, Karolinska Institutet
Other Study IDs: SAleman
Record Dates: First submitted 2017-06-21; First posted 2017-08-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C
Keywords: Sustained virological response; Whole genome sequencing
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Liver tissue from HCC and adjacent non-HCC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SVR and developed HCC: HCV patients with SVR and developed HCC plus available tissue from HCC

SUMMARY:
In this international collaboration study, the research group will analyze somatic mutations of hepatocellular carcinoma (HCC) developed after sustained virological response (SVR) in patients treated with hepatitis C (HCV) therapy

DETAILED DESCRIPTION:
Method Paired liver tissue samples will be collected from the tumour sections and also from the adjacent non-tumour tissues, for comparison in each individual. The tissues have been collected as part of routine clinical work/other studies, by liver biopsies or at liver resection/liver transplantation. Data regarding the patient characteristic will be collected. Whole genome sequencing analyses are planned to be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sustained virological response (SVR) after interferon (IFN)-containing or IFN-free treatment, and developed hepatocellular carcinoma (HCC)
* Available liver biopsies from hepatocellular carcinoma and non-HCC tissue

Exclusion Criteria:

* Co-infection with chronic hepatitis B (HBsAg positive) or HIV infection.
* Liver transplantation prior to treatment-start, leading to SVR.
* Patients with diagnosed HCC prior to treatment-start, leading to SVR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Please see eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Characterisation of genomic mutations of HCC, developed in HCV patients with SVR | 5 years
  Genetic characteristics of HCCs will be compared to non-HCC tissue

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bolinder, Prof, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual IPD will not be shared with other researchers